CLINICAL TRIAL: NCT05315011
Title: Evaluation of the Analgesic Effect of Cryotherapy in Anti-aromatase-induced Arthralgia: a Prospective Randomized Study
Brief Title: Assessment of Cryotherapy's Analgesic Impact in Anti-aromatase-induced Arthralgia
Acronym: CRYOMATASE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The cryotherapy center has closed due to liquidation.
Sponsor: University Hospital, Montpellier (Other)
Collaborators: CryoMed Millenaire (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RECHMPL20_0614; 2021-A02372-39 (Registry Identifier: ANSM register (ID-RCB))
Record Dates: First submitted 2022-03-29; First posted 2022-04-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Aromatase Inhibitors
Keywords: Aromatase Inhibitor; Arthralgias; Cryotherapy; Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Arthralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-body cryotherapy (Experimental): The exposure time will be 4 minutes and 30 seconds in -85°C.
  Interventions: Other: Whole-body cryotherapy
- Placebo cryotherapy (Placebo Comparator): The patient will be placed in a -85°C chamber for 1 minute as part of the placebo treatment.
  Interventions: Other: Placebo cryotherapy

INTERVENTIONS:
Other: Whole-body cryotherapy — The term "cryotherapy" refers to the process of chilling the body for medicinal purposes. WBC is carried out in a dedicated temperature and humidity controlled cryogenic chamber, which includes a brief exposure to extremely cold air. To avoid frostbite, only a few layers of clothes will be worn during the exposure. To avoid skin burns and necrosis, each participant must first remove their sweat before entering the cryochamber and a surgical mask is also worn to prevent moist air from being exhaled. Subjects will move their fingers and legs in the cryochamber and avoid holding their breath. The exposure time will be 4 minutes and 30 seconds in -85°C.
  Arms: Whole-body cryotherapy
Other: Placebo cryotherapy — The patient will be placed in a -85°C chamber for 1 minute as part of the placebo treatment.
  Arms: Placebo cryotherapy

SUMMARY:
The first aim of this comparative, randomized, prospective, multicenter study is to evaluate the analgesic effect at 6 weeks of whole-body cryotherapy, compared to placebo cryotherapy, in patients suffering from arthralgia under aromatase inhibitor treatment for hormone-dependent breast cancer in adjuvant situation.

The secondary objectives are to evaluate the tolerance of cryotherapy sessions and the evaluation of the impact of the cryotherapy sessions on the consumption of analgesics, the compliance of the treatment by anti-aromatases, the quality of life.

The patient and investigator will be blinded to the treatment. Only the cryotherapist will have knowledge of the treatment group:

* Whole Body Cryotherapy group (Arm A), or
* Placebo Cryotherapy group (Arm B). Patients consulting for the follow-up of a breast cancer and presenting arthralgias under anti-aromatase will be included in the study after verification of the inclusion and non-inclusion criteria and collection of consent.

The sessions will be performed according to the randomization arm as follows

* Whole body cryotherapy group: 10 sessions will be performed daily, over a period of 12 to 21 days. For each session, the patient enters a chamber at -85°C for 4 minutes 30 seconds.
* Placebo cryotherapy group: 10 sessions will be performed daily, over a period of 12 to 21 days. For each session, the patient enters a chamber at -85°C for 1 minute.

Each patient will complete the BPI-SF and HAQ questionnaires 15 days +/- 7 days prior to the start of cryotherapy, at the 6 week, 3 and 6 month post-cryotherapy visit.

Each patient will indicate the number of days of anti-aromatase therapy in the 6 months prior to inclusion and at 6 weeks, 3 and 6 months after cryotherapy. For this purpose, each patient will indicate the number of hormone therapy tablets taken in the 15 days prior to the inclusion visit, the 6 week, 3 and 6 month visit.

Each patient will indicate the analgesic treatments used, classified in three categories: levels 1, 2 and 3 at the inclusion consultation and at 6 weeks, 3 and 6 months after cryotherapy (analgesics taken during the 15 days preceding the visit).

The evaluation of the tolerance with the collection of the undesirable effects will be made before and at the end of each session by the professionals of the CryoMed. It will also be evaluated in the week following the end of cryotherapy during a telephone call.

DETAILED DESCRIPTION:
In 2018, the number of new cases of breast invasive cancer in France was estimated to be over 58 500, with a median age at diagnosis of 63 years.

The 5-year survival rate (as measured by age) has improved over time thanks to various treatments . Hormonotherapy is one of the disease's treatment options, and it includes a variety of molecules, including aromatase inhibitors. Despite their effectiveness, aromatase inhibitors cause a variety of side effects, including arthralgia in 35 percent to 50% of patients. The physiopathological mechanisms underlying these arthralgies would include articular inflammation, increased intra-articular fluid, and the appearance of a tenosynovitis. These side effects are frequently responsible for the premature discontinuation of hormone therapy and, as a result, the therapeutic effect of molecules. In order to improve the management of arthralgias caused by aromatase inhibitors, and because current recommendations are unclear, the effects of whole-body cryotherapy in patients who are taking an aromatase inhibitor for a hormono-dependent cancer in an adjuvant setting will be investigated. In fact, cryotherapy has already demonstrated its efficacy in the treatment of arthritic pain in a variety of diseases (rheumatoid arthritis,..).

This is a category 1, comparative, randomized, prospective, multicenter study. The patient and investigator will be blinded to the treatment. Only the cryotherapist will have knowledge of the treatment group.

Randomization will be performed after information and signature of informed consent on the day of the inclusion visit.

Patients will be randomized to either

* either in the Whole Body Cryotherapy group (Arm A),
* or in the placebo Cryotherapy group (Arm B). Randomization will be stratified by center, initial BPI score of most severe pain (greater than or equal to 7 vs. less than 7) and duration of initial pain exposure (greater than or equal to 6 months vs. less than 6 months). It will be centralized, accessible online (on the Internet) and programmed by minimization using the Ennov Clinical software (CSRandomization module) by the Clinical Research Unit of the Medical Information Department (DIM) of the Montpellier University Hospital. Patients will be recruited from the gynecological consultation service of the Arnaud de Villeneuve Hospital in Montpellier and the Caremeau Hospital in Nîmes. Patients consulting for the follow-up of a breast cancer and presenting arthralgias under anti-aromatase will be included in the study after verification of the inclusion and non-inclusion criteria and collection of consent.

Oral and written information will be given at the inclusion visit. Written consent will be collected at the end of the same visit after a reflection period.

Prior to the cryotherapy sessions, the patient will be asked not to exercise, take a shower or take any stimulant (tea or coffee) before a cryotherapy session. Before the first cryotherapy session, after a new verification of the absence of contraindication to cryotherapy, a blood pressure and temperature measurement will be taken (questionnaire before/after cryotherapy). The patient will receive information on the course of a cryotherapy session and will then be prepared: protection of recent skin wounds, wearing of a bathing suit and a surgeon's mask, protection of the extremities by gloves, slippers and a polar cap provided by the CryoMed.

Before each of the following sessions, a blood pressure reading and a skin temperature reading between the Achilles heel and the triceps will be taken. The occurrence of undesirable events since the last session will be investigated (questionnaire before/after cryotherapy).

After the patient enters the cryotherapy chamber (CryoAir, MecoTec), a permanent visual contact is kept on the patient throughout the session, thanks to a glass window. It is also possible to hear and communicate with the patient throughout the session.

The sessions will be performed according to the randomization arm as follows

* Whole body cryotherapy group: 10 sessions will be performed daily, over a period of 12 to 21 days. For each session, the patient enters a chamber at -85°C for 4 minutes 30 seconds.
* Placebo cryotherapy group: 10 sessions will be performed daily, over a period of 12 to 21 days. For each session, the patient enters a chamber at -85°C for 1 minute.

Patients can stop the cryotherapy session at any time. The duration of each session will be noted on the Before-After Cryotherapy questionnaire.

Finally, after the cyrotherapy sessions:

* Whole body cryotherapy group: In order to better understand the thermal shock and to adjust the following sessions, the patient's temperature will be recorded between her Achilles tendon and her triceps, as soon as she leaves the cryotherapy chamber:
* If > 12°C, the duration of exposure to -85°C will be increased by 20 seconds during the following sessions.
* If < 5°C, the duration of exposure to -85°C will be decreased by 20 seconds during the following sessions.

This process will be repeated with each new cryotherapy session.

• Placebo Cryotherapy Group: In order to promote blindness, the patient's temperature will be recorded between her Achilles tendon and her triceps, as soon as she leaves the cryotherapy chamber, but no change will be made to the duration of the following sessions.

Adverse events will be investigated at the end of each session (before/after cryotherapy questionnaire).

Each patient will complete the BPI-SF and HAQ questionnaires 15 days +/- 7 days prior to the start of cryotherapy, at the 6 week, 3 and 6 month post-cryotherapy visit.

Each patient will indicate the number of days of anti-aromatase therapy in the 6 months prior to inclusion and at 6 weeks, 3 and 6 months after cryotherapy. For this purpose, each patient will indicate the number of hormone therapy tablets taken in the 15 days prior to the inclusion visit, the 6 week, 3 and 6 month visit. A calendar will be given to each patient: the patient will indicate the use of hormone therapy and analgesics during the 15 days preceding the visits.

Each patient will indicate the analgesic treatments used, classified in three categories: levels 1, 2 and 3 at the inclusion consultation and at 6 weeks, 3 and 6 months after cryotherapy (analgesics taken during the 15 days preceding the visit).

The evaluation of the tolerance with the collection of the undesirable effects will be made before and at the end of each session by the professionals of the CryoMed. It will also be evaluated in the week following the end of cryotherapy during a telephone call.

A difference of 2 points or more in the BPI-SF score is considered as clinically significant. Under this assumption and that of a standard deviation of 2.3 points in both groups, the number of subjects to be analyzed to demonstrate a difference between the groups, with a two-sided alpha risk of 5% and a power of 80%, is 42 subjects, i.e. 21 subjects per group. In this study, there is a risk of attrition during or after the sessions, evaluated at 20%, and a risk of attrition of 20% between inclusion and the first session, due to organizational constraints and the possible appearance of contraindications to cryotherapy. In case of attrition between the inclusion and the first session, for a provisional reason, the patients could be re-included. A total of 70 inclusions are finally possible. As soon as 56 patients (28 per group) have completed at least one session, recruitment can be stopped.

The threshold of significance is set at 0.05 bilaterally for all analyses. Qualitative variables will be described by their number and percentage. Quantitative variables will be described by their mean, standard deviation, extrema, median and quartiles, in the randomized population, in the ITT population, in the PP population, in the safety population, and in each of the two groups within each of these populations. In addition, all baseline variables will be described in the included population. A flow-chart will be performed.

The main analysis will be performed in the ITT population by comparing the mean of the primary endpoint (most severe pain at 6 weeks) between the two groups by a test appropriate to the distribution of the data. Missing data will not be imputed.

The primary analysis will be supplemented by a secondary analysis of the YAC in which missing data will be imputed by multiple imputation, in the randomized population, and by an analysis in the PP population.

Secondary endpoints will be compared between the two groups, in the ITT population and in the PP population, without imputation for missing data:

* Mean comparisons for

  * Most severe pain at 3 and 6 months
  * BPI-SF composite pain severity and interference scores at 6 weeks, 3 and 6 months.
  * Health Assessment Questionnaire (HAQ) scores at 6 weeks, 3 and 6 months
  * Number of days on anti-aromatase therapy at 6 weeks, 3 and 6 months after cryotherapy.
* Comparison of percentages for the use of the different levels of analgesics at 6 weeks, 3 and 6 months.

Adverse events will be compared between the two groups in the safety population.

ELIGIBILITY:
Inclusion Criteria:

* Major non-menopausal patient
* Patient managed for histologically proven breast cancer
* Patient undergoing adjuvant anti-aromatase treatment (letrozole, anastrozole or exemestane) for at least 6 months
* Patient with arthralgias affecting one or more joints that have occurred or been exacerbated since the anti-aromatase treatment
* Patient with a score for the most severe pain experienced in the last week on the Brief Pain Inventory-Short Form (BPI-SF) ≥ 3.
* Patient with stable analgesic treatment for at least 15 days (without dose increase or change in step).

Exclusion Criteria:

* Infectious state
* Inflammatory, neurological or metabolic arthropathy
* Fracture or surgery of the painful extremity within the last 6 months
* Concomitant use of corticosteroid therapy
* Treatment with cryotherapy within 6 months prior to study inclusion
* Uncontrolled hypertension / Known coronary artery disease / History of myocardial infarction / History of cardiac rhythm disorder / Valvulopathy
* Pacemaker
* Previous venous thromboembolic event in progress
* Stage 3-4 arterial disease
* Unregulated hypothyroidism
* Severe Raynaud's syndrome
* Cryoglobulinemia
* Chronic respiratory insufficiency
* Polyneuropathy
* Acute renal or urinary pathology
* Epilepsy
* Alcohol and/or drug abuse
* Healing disorders
* Known allergy to cold
* Claustrophobia
* Uncontrolled hyperhydrosis
* Patient participating in another interventional research involving the human being
* Patient deprived of liberty by judicial or administrative decision.
* Patient protected by law under guardianship or curatorship
* Failure to obtain free, informed and written consent after a period of reflection
* Patient not affiliated or beneficiary of a national health insurance system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2027-05-04 (Estimated)

PRIMARY OUTCOMES:
The most intense pain | 2 weeks before the first cryotherapy session
  The most intense pain, on the Brief Pain Inventory Short Form (BPI-SF) at baseline (question 3 of BPI-SF).
  The two domains measured by the BPI-SF pain intensity (severity) and the impact of pain on functioning (interference). It is a pain and quality of life assessment measure used to examine pain intensity (sensory dimension) and functional impact (reactive dimension) in patients. Numerical scales from 0 to 10 indicate overall pain intensity, worst pain, least pain and current pain. A figure representing the human body is included to allow the patient to mark in which part of the body the pain is located.
The most intense pain | 6 weeks after the last cryotherapy session
  The most intense pain, on the Brief Pain Inventory Short Form (BPI-SF) The two domains measured by the BPI-SF pain intensity (severity) and the impact of pain on functioning (interference). It is a pain and quality of life assessment measure used to examine pain intensity (sensory dimension) and functional impact (reactive dimension) in patients. Numerical scales from 0 to 10 indicate overall pain intensity, worst pain, least pain and current pain. A figure representing the human body is included to allow the patient to mark in which part of the body the pain is located.

SECONDARY OUTCOMES:
The most intense pain | 3 months and 6 months after the last cryotherapy session
  The most intense pain, on the Brief Pain Inventory Short Form (BPI-SF)
Pain severity score | 6 weeks, 3 months, 6 months after the last cryotherapy session
  The BPI assesses pain severity at its "worst," "least," "average," and "now" (current pain) with the questions 3, 4, 5 and 6. Responses to these 4 items are rated from 0 (No pain) to 10 (Pain as bad as you can imagine). The average of these 4 items is the composite pain interference score.
Pain interference score | 6 weeks, 3 months, 6 months after the last cryotherapy session
  The question 9 of BPI-SF measures how much pain interfered with seven daily activities: general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. These 7 items are measured from 0 (Does not interference) to 10 (Completely interferes). BPI pain interference is scored as the mean of the seven interference items. This mean can be used if more than 50%, or four of seven, of the total items have been completed on a given administration.
HAQ score | 6 weeks, 3 months, 6 months after the last cryotherapy session
  The Health Assessment Questionnaire (HAQ) Each question is given the following score:
  0 = without any difficulty
  1. = with some difficulty
  2. = with great difficulty
  3. = unable to do so The rating for each of the 8 domains (dressing, body care, getting up, eating, walking, hygiene, catching, grasping, other activities) is the one corresponding to the highest score of the questions in that domain. If there is missing data for one or more questions in a particular domain, the rating is the highest score of the questions with an answer (missing data is not taken into account). The notion of the need for assistance from a third party and/or the use of devices can modify this scoring system. In this case the score for the domain concerned must be at least equal to 2 (a score of 3 is given if the highest score is equal to 3: in all other cases a score of 2 is given). The functional index is the sum of the scores of the various domains divided by the number of domains assessed (normally 8
Number of days of anti-aromatases taken during the 15 days preceding the visit | 6 weeks, 3 months, 6 months after the last cryotherapy session
  Number of days of taking anti-aromatase treatment at 6 weeks, 3 and 6 months after cryotherapy.
Number of analgesics | 6 weeks, 3 months, 6 months after the last cryotherapy session
  Use of analgesics taken during the 15 days preceding the visit classified into three categories: stage 1, 2 and 3, at 6 weeks, 3 and 6 months after cryotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Martha DURAES, MD, Principal Investigator — Montpellier University Hospital
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duraes M, Garbay M, Ferrer C, Duflos C, Rathat G. Effect of whole-body cryotherapy versus placebo cryotherapy on joint pain induced by aromatase inhibitors in women with early stage breast cancer: a randomised clinical trial. BMJ Open. 2023 Dec 9;13(12):e071756. doi: 10.1136/bmjopen-2023-071756. PMID 38070928